CLINICAL TRIAL: NCT07044414
Title: Effectiveness of Manual Acupuncture as an Adjuvant Therapy for Head and Neck Cancer Patients Undergoing Chemoradiation at the Radiation Oncology Polyclinic of RSUPN DR. Cipto Mangunkusumo
Brief Title: Effectiveness of Manual Acupuncture for Head and Neck Cancer Patients Undergoing Chemoradiation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Thia Wanudyo Hutami, Medical Doctor, Indonesia University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 25-06-0859
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-08

CONDITIONS: Head and Neck Neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: The intervention group will receive Manual Acupuncture, while the control group will receive sham Manual Acupuncture
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinding will be applied to participants and outcome assessors. Group allocation will not be disclosed to them to minimize assessment bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Manual Acupuncture
  Interventions: Device: Manual Acupuncture
- Control group (Sham Comparator): Sham Manual Acupuncture
  Interventions: Device: Sham Manual Acupuncture

INTERVENTIONS:
Device: Manual Acupuncture — Manual acupuncture is administered at bilateral ST36 Zusanli, SP6 Sanyinjiao, and midline points CV4 Guanyuan and CV6 Qihai using sterile, single-use 0.25 × 25 mm acupuncture needles. The insertion depth follows standard clinical practice and safety guidelines, with twirling stimulation performed at minutes 0 and 10. Each session lasts approximately 20 minutes and is conducted three times per week for a total of 21 sessions. Participants continue to receive their standard chemoradiotherapy for head and neck cancer.
  Arms: Intervention Group
Device: Sham Manual Acupuncture — Sham Manual acupuncture uses Park sham needles with telescopic tips that do not penetrate the skin, applied at the same acupoints (ST36, SP6, CV4, CV6) with identical procedure and appearance to mimic real acupuncture. Adhesive bases are used to fix the sham needles. Stimulation is mimicked at minutes 0 and 10. Sessions last the same duration and frequency as the intervention group. Participants also continue their standard chemoradiotherapy.
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to assess whether manual acupuncture (MA) is more effective than sham acupuncture in improving leukocyte count and reducing cancer-related fatigue (CRF) in head and neck cancer (HNC) patients undergoing chemoradiation therapy (CRT).

The main questions it aims to answer are:

* Does MA, compared to sham acupuncture, increase leukocyte and absolute neutrophil count (ANC) during CRT?
* Does MA, compared to sham acupuncture, reduce the severity of CRF as measured by the Visual Analogue Scale-Fatigue (VAS-F)?
* Does MA, compared to sham acupuncture, improve quality of life as measured by the EORTC QLQ-C30 questionnaire?

Participants will:

* Be adult patients with head and neck cancer who have completed induction chemotherapy and are undergoing CRT
* Be screened based on inclusion and exclusion criteria, including normal INR and platelet count above 25,000/mm³
* Be randomly assigned to either the MA group or sham group using Park sham needle
* Receive acupuncture at points ST36, SP6, CV4, and CV6 three times per week for seven sessions (total 21 sessions)
* Be evaluated for leukocyte count, ANC, fatigue (VAS-F), and quality of life (EORTC QLQ-C30) at baseline and at weekly intervals during therapy

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with head and neck cancer (HNC) based on histopathological examination, who have completed induction chemotherapy and are scheduled to undergo radiotherapy.
* Subjects aged ≥18 years.
* Subjects willing to participate in this study and provide written informed consent.
* Subjects with a Mini Mental State Examination (MMSE) score ≥24.
* Subjects with oxygen saturation ≥95% on room air.
* Subjects with stage III or IVA cancer.
* Subjects receiving a radiation dose of 66-70 Gy.

Exclusion Criteria:

* Subjects with severe comorbidities such as chronic kidney failure, metastatic liver cirrhosis, or heart disease.
* Subjects currently undergoing other therapies that may affect leukocyte counts, such as immunomodulatory therapy or high-dose corticosteroid use.
* Subjects who are still smoking or consuming alcohol.
* Subjects with blood clotting disorders or those currently taking anticoagulants, confirmed by laboratory results: neutrophils <1,000/mm³, platelets <25,000/mm³, INR >2.0, or partial thromboplastin time >20 seconds.
* Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-12-12 (Actual); Study Completion 2025-12-12 (Actual)

PRIMARY OUTCOMES:
Leukocyte Count | Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6 , Week 7
  Leukocyte count (cells/µL) will be measured through laboratory tests to evaluate changes in white blood cell levels.
Absolute Neutrophil Count (ANC) | Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6 , Week 7
  ANC (cells/µL) will be measured to assess neutrophil recovery and myelosuppression status.

SECONDARY OUTCOMES:
Visual Analogue Scale - Fatigue (VAS-F) | Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6 , Week 7
  Cancer-related fatigue will be assessed using the VAS-F scale ranging from 0 (no fatigue) to 10 (worst possible fatigue)
EORTC QLQ-C30 (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire) | Time Frame: Baseline, Week 7
  Quality of life will be measured using the EORTC QLQ-C30, a validated questionnaire with multiple domains (physical, emotional, role, social, cognitive function, and symptoms). Higher scores in global health reflect better QoL, while higher symptom scores indicate worse outcomes

CONTACTS AND LOCATIONS:
Overall Officials: KPEK FKUI-RSCM, Principal Investigator — The Health Research Ethics Commitee of Faculty Medicine
Locations (1):
- Universitas Indonesia, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided